CLINICAL TRIAL: NCT02310750
Title: A Phase 1, Within Cohort, Randomized, Double Blind, Third-party Open, Placebo-controlled, Single- And Multiple Dose Escalation, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06700841 In Healthy Subjects And Subjects With Plaque Psoriasis And Bioavailability Of A Tablet Formulation Relative To Suspension Formulation And The Effect Of Food On A Tablet Formulation Of Pf-06700841
Brief Title: A Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Study Of PF-06700841, With Bioavailability/Food Effect Investigation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: B7931001
Record Dates: First submitted 2014-11-18; First posted 2014-12-08 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — PF-06700841; Suspensions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-06700841 Oral Solution/Suspension (Experimental)
  Interventions: Drug: PF-06700841 oral solution/suspension
- PF-06700841 Tablet (Experimental)
  Interventions: Drug: PF-06700841 tablet
- Placebo (Placebo Comparator): Oral placebo comparator for the healthy subject single and multiple ascending dose periods, and the psoriasis multiple dose period. No placebo used for the bioavailability investigation.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06700841 oral solution/suspension — Oral solution or suspension of study drug PF-06700841 (once daily or twice daily during multiple dosing periods)
  Arms: PF-06700841 Oral Solution/Suspension
Other: Placebo — Matching placebo given during the single ascending and multiple dose periods
  Arms: Placebo
Drug: PF-06700841 tablet — PF-06700841 tablet formulation administered during the bioavailability / food effect investigation
  Arms: PF-06700841 Tablet

SUMMARY:
The main purpose of the study is to determine if PF-06700841 is safe and well tolerated when administered to humans. A secondary purpose is to assess what the body does to PF-06700841 and to assess what PF-06700841 does to the body when given as single and multiple doses. The pharmacokinetic properties of different forms of PF-06700841 may be studied (tablet and solution/suspension forms).

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria for Healthy Subject Cohorts:

* Healthy male subjects and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Key Inclusion Criteria for Psoriasis Subject Cohorts:

* Male subjects and/or female subjects of non-childbearing potential with a diagnosis of plaque psoriasis who are between the ages of 18 and 65 years, inclusive
* Have a diagnosis of plaque psoriasis for at least 6 months prior to first study dose

Exclusion Criteria:

Key Exclusion Criteria for Healthy Subject Cohorts:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Males of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product

Key Exclusion Criteria for Psoriasis Subject Cohorts:

* Currently have non plaque forms of psoriasis, (eg, erythrodermic, guttate, or pustular psoriasis).
* Have current drug induced psoriasis, eg, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, antimalarial drugs or lithium
* Males of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

REFERENCES:
- [Derived] Hughes JH, Qiu R, Banfield C, Dowty ME, Nicholas T. Population Pharmacokinetics of Oral Brepocitinib in Healthy Volunteers and Patients. Clin Pharmacol Drug Dev. 2022 Dec;11(12):1447-1456. doi: 10.1002/cpdd.1163. Epub 2022 Aug 31. PMID 36045513
- [Derived] Page KM, Suarez-Farinas M, Suprun M, Zhang W, Garcet S, Fuentes-Duculan J, Li X, Scaramozza M, Kieras E, Banfield C, Clark JD, Fensome A, Krueger JG, Peeva E. Molecular and Cellular Responses to the TYK2/JAK1 Inhibitor PF-06700841 Reveal Reduction of Skin Inflammation in Plaque Psoriasis. J Invest Dermatol. 2020 Aug;140(8):1546-1555.e4. doi: 10.1016/j.jid.2019.11.027. Epub 2020 Jan 21. PMID 31972249
- [Derived] Banfield C, Scaramozza M, Zhang W, Kieras E, Page KM, Fensome A, Vincent M, Dowty ME, Goteti K, Winkle PJ, Peeva E. The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a TYK2/JAK1 Inhibitor (PF-06700841) in Healthy Subjects and Patients With Plaque Psoriasis. J Clin Pharmacol. 2018 Apr;58(4):434-447. doi: 10.1002/jcph.1046. Epub 2017 Dec 21. PMID 29266308
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931001&StudyName=A%20Phase%201%2C%20Within%20Cohort%2C%20Randomized%2C%20Double%20Blind%2C%20Third-party%20Open%2C%20Placebo-controlled%2C%20Single-%20And%20Multiple%20Dose%20Escalation%2C%20Parallel%20Group%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Pf-06700841%20In%20Healthy%20Subjects%20And%20Subjects%20With%20Plaque%20Psoriasis%20And%20Bioavailability%20Of%20A%20Tablet%20Formulation%20Relative%20To%20Suspension%20Formulation%20And%20The%20Effect%20Of%20Food%20On%20A%20Tablet%20Formulation%20Of%20Pf-06700841

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study conducted in 7 Healthy Participant (HP) cohorts: 6 cohorts included Single Ascending Dose (SAD), 4 which continued into Multiple Ascending Dose (MAD) with washout, and a final cohort was tested for food effect (fasted/fed) with washout. 1 multiple dose (MD) cohort in Psoriasis subjects received drug at 2 different dose levels or placebo.
Groups:
- PF--06700841: 1 Milligram (mg) SAD Cohort: Healthy participants received PF-06700841 single tablet of 1 mg, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
- PF--06700841: 3 mg SAD Cohort: Healthy participants received PF-06700841 single tablet of 3 mg, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
- PF--06700841: 10 mg SAD Cohort Then MAD Cohort: Healthy participants received PF-06700841 single tablet of 10 mg, orally on Day 1 in the treatment period 1 for SAD cohort (8 days) followed by washout period of at least 7 days, then PF-06700841 tablet 10 mg orally, once daily from Day 1 to Day 10 in the treatment period 2 for MAD cohort (28 days).
- PF-06700841: 30 mg SAD Cohort Then MAD Cohort: Healthy participants received PF-06700841 single tablet of 30 mg, orally on Day 1 in the treatment period 1 for SAD cohort (8 days) followed by washout period of at least 7 days, then PF-06700841 tablet 30 mg orally, once daily from Day 1 to Day 10 in the treatment period 2 for MAD cohort (28 days).
- PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort: Healthy participants received PF-06700841 single tablet of 100 mg, orally on Day 1 in the treatment period 1 for SAD cohort (8 days) followed by washout period of at least 7 days, then PF-06700841 tablet 100 mg orally, once daily from Day 1 to Day 10 in the treatment period 2 for MAD cohort (28 days) followed by washout period of at least 7 days, then PF-06700841 tablet 50 mg orally, twice daily from Day 1 to Day 10 in the treatment period 3 for MAD cohort (28 days).
- PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort: Healthy participants received PF-06700841 single tablet of 200 mg, orally on Day 1 in the treatment period 1 for SAD cohort (8 days) followed by washout period of at least 7 days, then PF-06700841 tablet 175 mg orally, once daily from Day 1 to Day 10 in the treatment period 2 for MAD cohort (28 days).
- Placebo: SAD Cohort Then MAD Cohort: Healthy participants received placebo matched to PF-06700841 single tablet orally on Day 1 in the treatment period 1 for SAD cohort (8 days) followed by washout period of at least 7 days, then placebo matched to PF-06700841 tablet once daily from Day 1 to Day 10 in the treatment period 2 for MAD cohort (28 days) followed by washout period of at least 7 days followed by placebo matched to PF-06700841 tablet twice daily from Day 1 to Day 10 in the treatment period 3 for MAD cohort (28 days).
- Placebo: MAD Psoriasis Cohort: Participants with Psoriasis received placebo matched to PF-06700841 tablet orally, once daily from Day 1 to Day 28. Treatment period 2 for MAD Psoriasis cohort was of 56 days.
- PF-06700841: 30 mg MAD Psoriasis Cohort: Participants with Psoriasis received PF-06700841 tablet of 30 mg orally, once daily from Day 1 to Day 28. Treatment period 2 for MAD Psoriasis cohort was of 56 days.
- PF-06700841: 100 mg MAD Psoriasis Cohort: Participants with Psoriasis received PF-06700841 tablet of 100 mg orally, once daily from Day 1 to Day 28. Treatment period 2 for MAD Psoriasis cohort was of 56 days.
- PF-06700841: 100 mg Tablet Fasted, Tablet Fed, Solution Fasted: Participants received PF-06700841 100 mg tablet under fasted condition at Day 1 of treatment period 1 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fed condition at Day 1 of treatment period 2 (9 days) followed by second washout period (5 days) followed by PF-06700841 100 mg oral solution/suspension under fasted condition at Day 1 of treatment period 3 (9 days) in food effect cohorts.
- PF-06700841: 100 mg Solution Fasted, Tablet Fasted, Tablet Fed: Participants received PF-06700841 100 mg oral solution/suspension under fasted condition at Day 1 of treatment period 1 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fasted condition at Day 1 of treatment period 2 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fed condition at Day 1 of treatment period 3 (9 days) in food effect cohorts.
- PF-06700841: 100 mg Tablet Fed, Solution Fasted, Tablet Fasted: Participants received PF-06700841 100 mg tablet under fed condition at Day 1 of treatment period 1 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg oral solution/suspension under fasted condition at Day 1 of treatment period 2 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fasted condition at Day 1 of treatment period 3 (9 days) in food effect cohorts.
- PF-06700841: 100 mg Tablet Fasted, Solution Fasted, Tablet Fed: Participants received PF-06700841 100 mg tablet under fasted condition at Day 1 of treatment period 1 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg oral solution/suspension under fasted condition at Day 1 of treatment period 2 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fed condition at Day 1 of treatment period 3 (9 days) in food effect cohorts.
- PF-06700841: 100 mg Solution Fasted, Tablet Fed, Tablet Fasted: Participants received PF-06700841 100 mg oral solution/suspension under fasted condition at Day 1 of treatment period 1 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fed condition at Day 1 of treatment period 2 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fasted condition at Day 1 of treatment period 3 (9 days) in food effect cohorts.
- PF-06700841: 100 mg Tablet Fed, Tablet Fasted, Solution Fasted: Participants received PF-06700841 100 mg tablet under fed condition at Day 1 of treatment period 1 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg tablet under fasted condition at Day 1 of treatment period 2 (9 days) followed by washout period (5 days) followed by PF-06700841 100 mg oral solution/suspension under fasted condition at Day 1 of treatment period 3 (9 days) in food effect cohorts.
Period: HP Period 1
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF--06700841: 10 mg SAD Cohort Then MAD Cohort | PF-06700841: 30 mg SAD Cohort Then MAD Cohort | PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort | PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort | Placebo: SAD Cohort Then MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tablet Fasted, Tablet Fed, Solution Fasted | PF-06700841: 100 mg Solution Fasted, Tablet Fasted, Tablet Fed | PF-06700841: 100 mg Tablet Fed, Solution Fasted, Tablet Fasted | PF-06700841: 100 mg Tablet Fasted, Solution Fasted, Tablet Fed | PF-06700841: 100 mg Solution Fasted, Tablet Fed, Tablet Fasted | PF-06700841: 100 mg Tablet Fed, Tablet Fasted, Solution Fasted
Started | 7 | 6 | 6 | 6 | 8 | 8 | 13 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 6 | 6 | 6 | 5 | 8 | 8 | 12 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: HP Washout 1
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF--06700841: 10 mg SAD Cohort Then MAD Cohort | PF-06700841: 30 mg SAD Cohort Then MAD Cohort | PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort | PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort | Placebo: SAD Cohort Then MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tablet Fasted, Tablet Fed, Solution Fasted | PF-06700841: 100 mg Solution Fasted, Tablet Fasted, Tablet Fed | PF-06700841: 100 mg Tablet Fed, Solution Fasted, Tablet Fasted | PF-06700841: 100 mg Tablet Fasted, Solution Fasted, Tablet Fed | PF-06700841: 100 mg Solution Fasted, Tablet Fed, Tablet Fasted | PF-06700841: 100 mg Tablet Fed, Tablet Fasted, Solution Fasted
Started | 0 | 0 | 6 | 5 | 8 | 8 | 12 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 5 | 4 | 6 | 6 | 9 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: HP MAD, Psoriasis MD, HP Fasted/Fed
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF--06700841: 10 mg SAD Cohort Then MAD Cohort | PF-06700841: 30 mg SAD Cohort Then MAD Cohort | PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort | PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort | Placebo: SAD Cohort Then MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tablet Fasted, Tablet Fed, Solution Fasted | PF-06700841: 100 mg Solution Fasted, Tablet Fasted, Tablet Fed | PF-06700841: 100 mg Tablet Fed, Solution Fasted, Tablet Fasted | PF-06700841: 100 mg Tablet Fasted, Solution Fasted, Tablet Fed | PF-06700841: 100 mg Solution Fasted, Tablet Fed, Tablet Fasted | PF-06700841: 100 mg Tablet Fed, Tablet Fasted, Solution Fasted
Started | 0 | 0 | 5 | 4 | 6 | 6 | 9 | 9 | 14 | 7 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 5 | 3 | 6 | 4 | 9 | 7 | 6 | 4 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 8 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: HP Washout 2
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF--06700841: 10 mg SAD Cohort Then MAD Cohort | PF-06700841: 30 mg SAD Cohort Then MAD Cohort | PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort | PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort | Placebo: SAD Cohort Then MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tablet Fasted, Tablet Fed, Solution Fasted | PF-06700841: 100 mg Solution Fasted, Tablet Fasted, Tablet Fed | PF-06700841: 100 mg Tablet Fed, Solution Fasted, Tablet Fasted | PF-06700841: 100 mg Tablet Fasted, Solution Fasted, Tablet Fed | PF-06700841: 100 mg Solution Fasted, Tablet Fed, Tablet Fasted | PF-06700841: 100 mg Tablet Fed, Tablet Fasted, Solution Fasted
Started | 0 | 0 | 0 | 0 | 6 | 0 | 9 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: HP MAD and Fasted/Fed
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF--06700841: 10 mg SAD Cohort Then MAD Cohort | PF-06700841: 30 mg SAD Cohort Then MAD Cohort | PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort | PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort | Placebo: SAD Cohort Then MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tablet Fasted, Tablet Fed, Solution Fasted | PF-06700841: 100 mg Solution Fasted, Tablet Fasted, Tablet Fed | PF-06700841: 100 mg Tablet Fed, Solution Fasted, Tablet Fasted | PF-06700841: 100 mg Tablet Fasted, Solution Fasted, Tablet Fed | PF-06700841: 100 mg Solution Fasted, Tablet Fed, Tablet Fasted | PF-06700841: 100 mg Tablet Fed, Tablet Fasted, Solution Fasted
Started | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-06700841: 100 mg Food Effect Cohort: All participants who received either PF-06700841 100 mg tablet under fasted condition or PF-06700841 100 mg tablet under fed condition or PF-06700841 100 mg oral solution/suspension under fasted condition in either 1 of the 3 treatment period in any 1 of the 6 treatment sequences in food effects cohort of the study.
- Total: Total of all reporting groups
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF--06700841: 10 mg SAD Cohort Then MAD Cohort | PF-06700841: 30 mg SAD Cohort Then MAD Cohort | PF--06700841: 100 mg SAD, 100 mg MAD, 50 mg MAD Cohort | PF--06700841: 200 mg SAD Cohort, 175 mg MAD Cohort | Placebo: SAD Cohort Then MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Food Effect Cohort | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 8 | 8 | 13 | 9 | 14 | 7 | 12 | 96
Age, Customized [Number; unit: participants]
  18-44 Years | 4 | 2 | 1 | 4 | 5 | 6 | 11 | 6 | 6 | 5 | 5 | 55
  45-64 Years | 3 | 4 | 5 | 2 | 3 | 2 | 2 | 3 | 8 | 2 | 7 | 41
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 6
  Male | 7 | 6 | 6 | 6 | 8 | 7 | 12 | 8 | 12 | 7 | 11 | 90

OUTCOME MEASURES:

1. Primary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Blood Pressure at Day 1
Time Frame: Baseline, 24 hours post-dose on Day 1
Population: Full analysis set (FAS) included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Groups:
- Placebo: SAD Cohort: Healthy participants received single tablet of placebo matched to PF-06700841, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
- PF-06700841: 10 mg SAD Cohort: Healthy participants received PF-06700841 single tablet of 10 mg, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
- PF-06700841: 30 mg SAD Cohort: Healthy participants received PF-06700841 single tablet of 30 mg, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
- PF-06700841: 100 mg SAD Cohort: Healthy participants received PF-06700841 single tablet of 100 mg, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
- PF-06700841: 200 mg SAD Cohort: Healthy participants received PF-06700841 single tablet of 200 mg, orally on Day 1. Treatment period 1 for SAD cohort was of 8 days.
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
millimeter of mercury (mmHg)
  Supine Systolic Blood Pressure (SBP): Baseline | 114.2 (11.97) | 110.6 (6.70) | 108.7 (7.76) | 102.8 (6.62) | 117.8 (9.54) | 112.4 (12.26) | 115.3 (5.99)
  Supine SBP: Change at Day 1 | -2.6 (6.40) | -8.1 (9.32) | 1.0 (8.17) | 9.5 (5.96) | -1.5 (4.64) | 2.1 (11.28) | -5.3 (7.91)
  Supine Diastolic blood pressure (DBP): Baseline | 64.0 (8.55) | 67.0 (8.77) | 66.2 (8.42) | 58.7 (8.19) | 70.3 (7.39) | 66.9 (8.98) | 70.5 (5.88)
  Supine DBP: Change at Day 1 | -1.1 (7.44) | -5.3 (9.05) | 2.2 (9.56) | 4.7 (715) | 2.5 (8.83) | -0.1 (8.36) | -2.3 (6.14)

2. Primary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Blood Pressure at Day 10
Time Frame: Baseline, 16 hours post-dose on Day 10
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Once Daily MAD Cohort: Healthy participants received placebo matched to PF-06700841 tablet orally once daily from Day 1 to Day 10. Treatment period 2 for MAD cohort was of 28 days.
- Placebo: Twice Daily MAD Cohort: Healthy participants received placebo matched to PF-06700841 tablet orally twice daily from Day 1 to Day 10. Treatment period 3 for MAD cohort was of 28 days.
- PF-06700841: 10 mg Once Daily MAD Cohort: Healthy participants received PF-06700841 tablet of 10 mg orally, once daily from Day 1 to Day 10. Treatment period 2 for MAD period was of 28 days.
- PF-06700841: 30 mg Once Daily MAD Cohort: Healthy participants received PF-06700841 tablet of 30 mg orally, once daily from Day 1 to Day 10. Treatment period 2 for MAD period was of 28 days.
- PF-06700841: 100 mg Once Daily MAD Cohort: Healthy participants received PF-06700841 tablet of 100 mg orally, once daily from Day 1 to Day 10. Treatment period 2 for MAD period was of 28 days.
- PF-06700841: 50 mg Twice Daily MAD Cohort: Healthy participants received PF-06700841 tablet of 50 mg orally, twice daily from Day 1 to Day 10. Treatment period 3 for MAD cohort was of 28 days.
- PF-06700841: 175 mg Once Daily MAD Cohort: Healthy participants received PF-06700841 tablet of 175 mg orally, once daily from Day 1 to Day 10. Treatment period 2 for MAD period was of 28 days.
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
mmHg
  Supine SBP: Baseline (n=9,2,5,4,6,5,6) | 112.2 (9.78) | 106.5 (3.54) | 103.6 (7.64) | 110.3 (5.19) | 111.5 (13.35) | 108.6 (18.45) | 115.8 (8.66)
  Supine SBP: Change at Day 10 (n=9,2,5,3,6,4,4) | 4.0 (9.12) | 12.5 (2.12) | -0.2 (7.69) | 8.7 (10.69) | 7.7 (12.97) | -3.5 (8.89) | -5.3 (4.86)
  Supine DBP: Baseline (n=9,2,5,4,6,5,6) | 60.3 (4.15) | 61.5 (7.78) | 56.2 (4.02) | 65.5 (3.70) | 68.8 (9.06) | 59.2 (16.80) | 66.2 (8.06)
  Supine DBP: Change at Day 10 (n=9,2,5,3,6,4,4) | 4.2 (7.26) | 6.0 (4.24) | 2.2 (6.76) | 5.7 (1.53) | 3.2 (9.62) | -4.3 (9.14) | 2.0 (5.48)

3. Primary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Blood Pressure at Day 28
Time Frame: Baseline, 16 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
mmHg
  Supine SBP: Baseline (n =9, 14, 7) | 115.0 (13.21) | 120.1 (10.91) | 112.9 (8.11)
  Supine SBP: Change at Day 28 (n =8, 7, 5) | -5.3 (11.87) | -8.9 (9.94) | 1.0 (11.94)
  Supine DBP: Baseline (n =9, 14, 7) | 67.8 (7.93) | 69.9 (7.94) | 66.6 (7.55)
  Supine DBP: Change at Day 28 (n =8, 7, 5) | -3.9 (5.51) | -7.0 (6.00) | -0.8 (16.96)

4. Primary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Pulse Rate at Day 1
Time Frame: Baseline, 24 hours post-dose on Day 1
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
beats per minute (bpm)
  Baseline | 57.5 (6.36) | 68.6 (13.81) | 67.2 (9.66) | 56.0 (8.05) | 67.3 (9.24) | 55.8 (11.77) | 57.8 (6.54)
  Change at Day 1 | 1.0 (3.42) | 6.1 (7.58) | 2.5 (6.28) | 3.0 (8.10) | 0.7 (5.54) | -1.1 (3.94) | 2.6 (6.39)

5. Primary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Pulse Rate at Day 10
Time Frame: Baseline, 16 hours post-dose on Day 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
bpm
  Baseline (n =9,2,5,4,6,5,6) | 59.3 (12.58) | 59.0 (1.41) | 55.8 (7.36) | 60.8 (4.99) | 61.5 (7.50) | 66.0 (9.43) | 60.5 (9.61)
  Change at Week 10 (n =9,2,5,3,6,4,4,) | -2.3 (12.21) | -0.5 (0.71) | -1.6 (5.18) | -4.0 (7.21) | -6.3 (8.24) | -2.5 (4.43) | -1.0 (6.38)

6. Primary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Pulse Rate at Day 28
Time Frame: Baseline, 16 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
bpm
  Baseline (n =9, 14, 7) | 61.8 (8.07) | 61.4 (9.52) | 64.9 (6.04)
  Change at Week 28 (n =8, 7, 5) | -1.9 (5.38) | -5.3 (7.41) | -3.0 (3.39)

7. Primary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Oral Temperature at Day 1
Time Frame: Baseline, 24 hours post-dose on Day 1
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
degree celsius
  Baseline | 36.79 (0.155) | 36.83 (0.359) | 36.65 (0.187) | 36.82 (0.194) | 36.80 (0.141) | 36.69 (0.164) | 36.63 (0.149)
  Change at Day 1 | 0.05 (0.151) | -0.11 (0.418) | 0.35 (0.281) | 0.05 (0.235) | 0.07 (0.103) | -0.03 (0.238) | 0.05 (0.177)

8. Primary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Oral Temperature at Day 10
Time Frame: Baseline, 16 hours post-dose on Day 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
degree celsius
  Baseline (n =9, 2, 5, 4, 6, 5, 6) | 36.71 (0.136) | 36.70 (0.141) | 36.76 (0.182) | 36.68 (0.126) | 36.83 (0.163) | 36.76 (0.167) | 36.75 (0.235)
  Change at Day 10 (n =9, 2, 5, 3, 6, 4, 4) | 0.08 (0.228) | 0.05 (0.071) | -0.22 (0.164) | -0.10 (0.100) | -0.22 (0.214) | -0.17 (0.206) | 0.05 (0.208)

9. Primary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Oral Temperature at Day 28
Time Frame: Baseline, 16 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees celsius
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
degrees celsius
  Baseline (n = 9, 14, 7) | 36.74 (0.151) | 36.67 (0.213) | 36.80 (0.277)
  Change at Week 28 (n= 8, 7, 5) | 0.01 (0.223) | -0.04 (0.369) | -0.20 (0.300)

10. Primary Outcome: Number of Participants With Change From Baseline in Physical Examinations
Description: Physical examinations included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems.
Time Frame: SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 28, MAD Psoriasis Cohort: Baseline up to Day 56, Food Effect Cohort: Baseline up to Day 37
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- PF-06700841: 100 mg Tab Fasted (Food Effect Cohort): All participants who received PF-06700841 100 mg tablet under fasted condition in either 1 of the 3 treatment period in food effects cohort of the study.
- PF-06700841: 100 mg Solution Fasted (Food Effect Cohort): All participants who received PF-06700841 100 mg oral solution/suspension under fasted condition in either 1 of the 3 treatment period in food effects cohort of the study.
- PF-06700841: 100 mg Tablet Fed (Food Effect Cohort): All participants who received PF-06700841 100 mg tablet under fed condition in either 1 of the 3 treatment period in food effects cohort of the study.
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8 | 9 | 2 | 5 | 4 | 6 | 5 | 6 | 9 | 14 | 7 | 12 | 12 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0

11. Primary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) at Day 1
Time Frame: Baseline, 24 hours post-dose on Day 1
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
millisecond (msec)
  PR Interval: Baseline | 175.7 (14.52) | 149.7 (18.62) | 163.1 (13.58) | 168.2 (14.63) | 163.6 (19.37) | 175.8 (18.86) | 165.9 (7.65)
  PR Interval: Change at Day 1 | -0.9 (6.78) | 6.7 (8.12) | -2.4 (6.65) | 2.2 (5.45) | -2.1 (5.95) | 3.3 (5.62) | 0.5 (7.54)
  QRS Complex: Baseline | 97.7 (15.40) | 92.9 (9.30) | 97.4 (10.43) | 102.9 (8.74) | 99.8 (14.61) | 101.7 (6.87) | 92.0 (5.81)
  QRS Complex: Change at Day 1 | -3.1 (12.73) | -1.5 (5.98) | -2.2 (4.06) | -1.7 (3.55) | -2.9 (3.45) | -2.0 (5.19) | 1.7 (2.33)
  QT Interval: Baseline | 408.4 (21.42) | 374.0 (21.81) | 384.3 (26.20) | 404.2 (19.89) | 387.5 (12.0) | 421.3 (29.94) | 407.1 (20.71)
  QT Interval: Change at Day 1 | -5.9 (10.41) | -3.8 (10.21) | -3.1 (9.43) | -8.2 (9.25) | -0.8 (4.56) | -0.8 (11.61) | -3.3 (14.78)
  QTC Interval: Baseline | 397.7 (16.51) | 390.9 (20.95) | 400.6 (11.90) | 392.2 (13.42) | 402.7 (20.69) | 400.0 (7.60) | 402.7 (14.10)
  QTC Interval: Change at Day 1 | -0.2 (9.24) | -2.3 (5.45) | -1.9 (7.61) | 2.4 (9.42) | -4.6 (4.41) | 4.2 (7.75) | 3.2 (5.76)

12. Primary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) at Day 10
Time Frame: Baseline, 16 hours post-dose on Day 10
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
msec
  PR Interval: Baseline (n =9,2,5,4,6,5,6) | 176.9 (16.31) | 180.0 (1.41) | 167.6 (10.69) | 169.0 (22.38) | 168.5 (18.79) | 171.6 (14.77) | 168.0 (6.66)
  PR Interval: Change at Day 10 (n =9,2,5,3,6,4,4) | 5.2 (3.59) | 4.7 (6.60) | 7.7 (5.36) | 14.3 (8.41) | 7.3 (10.07) | 11.2 (5.14) | 1.4 (2.33)
  QRS Complex: Baseline (n =9,2,5,4,6,5,6) | 96.6 (5.83) | 96.0 (7.07) | 103.0 (9.14) | 101.0 (20.05) | 102.7 (8.52) | 103.0 (8.34) | 95.2 (8.70)
  QRS Complex: Change at Day 10 (n =9,2,5,3,6,4,4) | 0.9 (1.60) | -0.5 (6.36) | -3.2 (9.49) | -2.3 (6.17) | 1.3 (5.32) | 2.9 (5.26) | -1.7 (1.83)
  QT Interval: Baseline (n =9,2,5,4,6,5,6) | 411.9 (27.98) | 425.5 (10.61) | 407.4 (18.17) | 398.0 (9.56) | 399.7 (16.12) | 397.0 (23.29) | 401.8 (27.66)
  QT Interval: Change at Day 10 (n =9,2,5,3,6,4,4) | -3.9 (14.72) | 1.0 (11.79) | -1.0 (23.42) | 2.6 (9.26) | 1.3 (16.66) | 2.3 (5.51) | 2.1 (23.19)
  QTC Interval: Baseline (n =9,2,5,4,6,5,6) | 398.7 (11.35) | 415.5 (4.95) | 396.4 (15.53) | 401.5 (15.37) | 396.0 (6.54) | 403.2 (6.26) | 403.5 (11.96)
  QTC Interval: Change at Day 10 (n =9,2,5,3,6,4,4) | -0.3 (9.82) | -1.5 (10.14) | -2.9 (3.00) | -5.0 (10.49) | -1.3 (10.34) | -0.3 (4.46) | 2.0 (10.47)

13. Primary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) at Day 28
Time Frame: Baseline, 16 hours post-dose on Day 28
Population: FAS included all participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
msec
  PR Interval: Baseline (n =9, 14, 7) | 169.4 (15.26) | 156.1 (17.78) | 154.7 (11.51)
  PR Interval: Change at Day 28 (n =8, 7, 5) | -0.6 (10.19) | 11.1 (5.95) | 4.1 (7.09)
  QRS Complex: Baseline (n =9, 14, 7) | 100.6 (8.32) | 97.4 (10.27) | 93.0 (5.87)
  QRS Complex: Change at Day 28 (n= 8, 7, 5) | 0.5 (4.86) | 0.8 (4.73) | 3.8 (5.26)
  QT Interval: Baseline (n =9, 14, 7) | 404.4 (17.48) | 411.6 (31.01) | 379.0 (18.94)
  QT Interval: Change at Day 28 (n =8, 7, 5) | -17.9 (16.00) | -22.6 (23.04) | -5.3 (9.43)
  QTC Interval: Baseline (n=9, 14, 7) | 409.7 (14.46) | 409.0 (14.92) | 392.0 (19.04)
  QTC Interval: Change at Day 28 (n= 8, 7, 5) | -8.7 (10.83) | -9.6 (7.89) | -2.7 (13.18)

14. Primary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Heart Rate at Day 1
Time Frame: Baseline, 24 hours post-dose on Day 1
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
bpm
  Baseline | 56.1 (6.83) | 70.3 (16.46) | 69.2 (12.06) | 55.3 (5.65) | 67.7 (8.82) | 53.0 (8.92) | 58.0 (5.17)
  Change at Day 1 | 2.2 (3.74) | 1.6 (2.81) | 0.3 (3.27) | 4.6 (4.64) | -2.3 (1.72) | 2.0 (3.19) | 3.4 (5.79)

15. Primary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Heart Rate at Day 10
Time Frame: Baseline, 16 hours post-dose on Day 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
bpm
  Baseline (n =9, 2, 5, 4, 6, 5, 6) | 55.1 (7.15) | 55.5 (2.12) | 55.4 (4.45) | 61.0 (2.94) | 58.5 (6.38) | 63.0 (7.38) | 61.2 (7.96)
  Change at Day 10 (n = 9, 2, 5, 3, 6, 4, 4) | -1.2 (10.33) | 7.7 (6.13) | -1.1 (7.22) | -3.0 (4.04) | -2.3 (5.12) | -1.8 (5.79) | -1.3 (4.04)

16. Primary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Heart Rate at Day 28
Time Frame: Baseline, 16 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
bpm
  Baseline (n =9, 14, 7) | 63.1 (9.15) | 60.2 (11.25) | 66.0 (4.93)
  Change at Day 28 (n =8, 7, 5) | 5.2 (5.28) | 4.0 (8.73) | 1.4 (5.60)

17. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation Due to AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug up to the end of study (up to Day 8 in SAD cohort, Day 28 in MAD cohort, Day 56 in MAD Psoriasis cohort, Day 37 in Food effect cohort), that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAE and non-SAE.
Time Frame: as for outcome 10
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8 | 9 | 2 | 5 | 4 | 6 | 5 | 6 | 9 | 14 | 7 | 12 | 12 | 12
participants
  AEs | 2 | 1 | 1 | 0 | 1 | 3 | 2 | 0 | 1 | 3 | 2 | 3 | 5 | 5 | 5 | 11 | 6 | 1 | 2 | 0
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Withdrawal due to AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0

18. Primary Outcome: Number of Adverse Events (AEs) According to Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs were classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.
Time Frame: as for outcome 10
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: adverse events
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8 | 9 | 2 | 5 | 4 | 6 | 5 | 6 | 9 | 14 | 7 | 12 | 12 | 12
adverse events
  Mild | 2 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 3 | 2 | 2 | 6 | 6 | 7 | 16 | 16 | 1 | 2 | 0
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for abnormality:hematology: hemoglobin, hematocrit, red blood cell count: less than(<) 0.8*lower limit of normal (LLN); mean corpuscular volume; mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration: <0.9*LLN,>1.1*upper limit of normal (ULN); platelets: <0.5*LLN,>1.75*ULN, white blood cell count: <0.6*LLN, >1.5*ULN; lymphocytes, total neutrophils: <0.8*LLN, >1.2*ULN; eosinophils, basophils, monocytes: >1.2*ULN; coagulation: activated partial thromboplastin time, prothrombin, prothrombin international ratio: >1.1*ULN; liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN; renal function:blood urea nitrogen,creatinine: >1.3*ULN; uric acid: >1.2*ULN; electrolytes: sodium, potassium, chloride, calcium, bicarbonate: <0.9*LLN,>1.1*ULN; urinalysis: pH<4.5, >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite; Other(glucose: <0.6*LLN,>1.5*ULN)
Time Frame: as for outcome 10
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8 | 9 | 2 | 5 | 4 | 6 | 5 | 6 | 9 | 14 | 7 | 12 | 12 | 12
participants | 7 | 4 | 4 | 6 | 6 | 6 | 7 | 6 | 0 | 5 | 4 | 6 | 5 | 6 | 7 | 13 | 7 | 5 | 1 | 3

20. Primary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Creatinine Clearance at Day 1
Description: Creatinine clearance is a measure of kidney function. Creatinine clearance is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time.
Time Frame: Baseline, 24 hours post-dose on Day 1
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: milliliter per minute (mL/min)
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 12 | 7 | 6 | 6 | 5 | 8 | 8
milliliter per minute (mL/min)
  Baseline | 117.7 (28.70) | 93.0 (36.60) | 133.8 (29.76) | 95.8 (53.07) | 117.0 (28.70) | 129.6 (25.43) | 114.4 (24.64)
  Change at Day 1 | 24.3 (63.75) | -0.4 (35.35) | -2.7 (11.27) | 15.8 (36.79) | -6.4 (6.35) | -17.6 (28.67) | 73.4 (227.50)

21. Primary Outcome: Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Change From Baseline in Creatinine Clearance at Day 10
Description: as for outcome 20
Time Frame: Baseline, 16 hours post-dose on Day 10
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6 | 9 | 14 | 7
mL/min
  Baseline (n =9, 2, 5, 4, 6, 5, 6, 2, 2, 7) | 114.4 (27.75) | 111.0 (1.41) | 112.6 (42.08) | 115.0 (34.13) | 142.5 (56.68) | 138.4 (51.27) | 83.0 (39.73) | 140.5 (55.86) | 158.0 (36.77) | 172.4 (51.74)
  Change at Day 10 (n =9, 2, 5, 3, 6, 4, 4, 2, 2, 7) | 0.7 (33.29) | -2.5 (57.28) | 26.8 (46.90) | -19.0 (25.51) | -47.0 (55.68) | -39.5 (29.86) | 3.5 (40.42) | -38.5 (60.10) | -50.0 (4.24) | -67.3 (61.45)

22. Primary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Creatinine Clearance at Day 28
Description: as for outcome 20
Time Frame: Baseline, 16 hours post-dose on Day 28
Population: FAS included all participants who were randomized to treatment and received at least 1 dose of study medication. Here, 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 1 | 2 | 5
mL/min | -10.0 (0.0) | -35.0 (33.94) | -67.6 (50.33)

23. Primary Outcome: Food Effect Cohort: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06700841
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post dose on Day 1
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 12 | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 6463 (46) | 6720 (43) | 5321 (53)

24. Primary Outcome: Food Effect Cohort: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06700841
Description: Area under the plasma concentration time-curve from time zero to the time of last measured concentration (AUClast).
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post dose on Day 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 12 | 12 | 12
ng*hr/mL | 6447 (46) | 6694 (43) | 5305 (53)

25. Primary Outcome: Food Effect Cohort: Maximum Observed Plasma Concentration (Cmax) of PF-06700841
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post dose on Day 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 12 | 12 | 12
nanogram per milliliter (ng/mL) | 1022 (35) | 1084 (40) | 656.6 (26)

26. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Maximum Observed Plasma Concentration (Cmax) of PF-06700841
Time Frame: SAD: pre-dose, 0.5,1,2,4,6,8,12,16,24,36,48,72,96 hour post dose on Day 1; MAD: pre-dose 0.5,1,2,4,6,8,12,24 hour post-dose on Day 10; MAD Psoriasis: pre-dose, 0.5,1,2,4,6,8,12,16,24 hours post dose on Day 28
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of interest. Here, 'N' signifies those participants who were evaluable for this outcome measure. Data for this outcome was not planned to be analyzed for Placebo: SAD Cohort, MAD Cohort, MAD Psoriasis Cohort arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 8 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5
ng/mL | 5.138 (52) | 18.21 (92) | 79.30 (35) | 271.3 (21) | 748.4 (35) | 2460 (37) | 63.42 (11) | 286.6 (17) | 734.1 (29) | 522.0 (31) | 2091 (28) | 204.7 (43) | 924.2 (13)

27. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06700841
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Median (Full Range); unit: hour
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 8 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5
hour | 1.00 [0.500 to 2.00] | 1.00 [0.500 to 1.00] | 0.500 [0.500 to 1.00] | 1.00 [0.500 to 1.02] | 1.00 [0.500 to 2.00] | 1.00 [0.500 to 2.00] | 1.00 [1.00 to 1.03] | 1.00 [1.00 to 1.00] | 1.50 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 0.984 [0.500 to 2.00] | 1.00 [0.983 to 1.00] | 2.00 [1.00 to 2.00]

28. Secondary Outcome: Food Effect Cohort: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF--06700841
Time Frame: Pre--dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post dose on Day 1
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 12 | 12 | 12
hour | 0.500 (0.500) [0.500 to 2.00] | 1.00 (1.2965) [0.500 to 2.00] | 4.00 (1.4383) [1.00 to 4.00]

29. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06700841
Description: as for outcome 23
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post dose on Day 1
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of interest. Here, 'N' signifies those participants who were evaluable for this outcome measure. Data for this outcome was not planned to be analyzed for Placebo: SAD Cohort arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 7 | 8
ng*hr/mL | NA (NA) [0.500 to 2.00] — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 145.8 (61) [0.500 to 1.00] | 353.8 (31) [0.500 to 1.00] | 1439 (65) [0.500 to 1.02] | 4797 (62) [0.500 to 2.00] | 18410 (46) [0.500 to 2.00]

30. Secondary Outcome: Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06700841
Description: Area under the plasma concentration versus time curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 24 hours for MAD once daily cohorts, 12 hours for MAD twice daily cohort and 24 hours for MAD Psoriasis cohort.
Time Frame: MAD: pre-dose 0.5, 1, 2, 4, 6, 8, 12, 24 hour post-dose on Day 10; MAD Psoriasis: pre-dose, 0.5,1,2,4,6,8,12,16,24 hours post dose on Day 28
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of interest. Here, 'N' signifies those participants who were evaluable for this outcome measure. Data for this outcome was not planned to be analyzed for Placebo: MAD Cohort, MAD Psoriasis Cohort arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 5 | 3 | 6 | 4 | 4 | 7 | 5
ng*hr/mL | 422.8 (41) | 1880 (52) | 6089 (38) | 3560 (35) | 16180 (15) | 990.0 (103) | 7672 (43)

31. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06700841
Description: Area under the plasma concentration time-curve from time zero to the time of last measured concentration (AUClast).
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post dose on Day 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8
ng*hr/mL | 17.71 (114) [0.500 to 2.00] | 79.18 (239) [0.500 to 1.00] | 340.4 (30) [0.500 to 1.00] | 1431 (65) [0.500 to 1.02] | 5041 (59) [0.500 to 2.00] | 18400 (46) [0.500 to 2.00]

32. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) of PF-06700841
Description: Dose normalized (dn) Cmax was calculated by dividing Cmax by the exact dose of PF 06700841 (in mg) administered to a participant.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram/milliliter]/milligram
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 8 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5
[nanogram/milliliter]/milligram | 5.138 (52) | 6.061 (92) | 7.930 (35) | 9.033 (21) | 7.484 (35) | 12.31 (37) | 6.342 (11) | 9.563 (17) | 7.341 (29) | 10.43 (30) | 11.97 (28) | 6.827 (43) | 9.242 (13)

33. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Dose Normalized Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf[dn]) of PF-06700841
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUCinf(dn) was calculated by dividing AUCinf by the exact dose of PF-06700841 (in mg) administered to a participant.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post dose on Day 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram*hour/milliliter]/milligram
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 7 | 8
[nanogram*hour/milliliter]/milligram | NA (NA) [0.500 to 2.00] — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 48.65 (61) [0.500 to 1.00] | 35.38 (31) [0.500 to 1.00] | 47.97 (65) [0.500 to 1.02] | 47.97 (62) [0.500 to 2.00] | 92.13 (46) [0.500 to 2.00]

34. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast[dn]) of PF-06700841
Description: Area under the plasma concentration time-curve from time zero to the time of last measured concentration (AUClast). AUClast(dn) was calculated by dividing AUClast by the exact dose of of PF-06700841 (in mg) administered to a participant.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post dose on Day 1
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng*hr/mL]/mg
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8
[ng*hr/mL]/mg | 17.71 (114) [0.500 to 2.00] | 26.38 (239) [0.500 to 1.00] | 34.04 (30) [0.500 to 1.00] | 47.64 (65) [0.500 to 1.02] | 50.41 (59) [0.500 to 2.00] | 92.09 (46) [0.500 to 2.00]

35. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Dose Normalized Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau[dn]) of PF-06700841
Description: Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 24 hours for MAD once daily cohorts, 12 hours for MAD twice daily cohort. AUCtau(dn) was calculated by dividing AUCtau by the exact dose of of PF-06700841 (in mg) administered to a participant.
Time Frame: pre-dose 0.5,1,2,4,6,8,12,24 hour post-dose on Day 10
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of interest. Here, 'N' signifies those participants who were evaluable for this outcome measure. Data for this outcome was not planned to be analyzed for Placebo Once Daily and Twice Daily: MAD Cohort arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng*hr/mL]/mg
Arm/Group | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 5 | 3 | 6 | 4 | 4
[ng*hr/mL]/mg | 42.28 (41) | 62.68 (51) | 60.89 (38) | 71.15 (36) | 92.30 (16)

36. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Plasma Decay Half-Life (t1/2) of PF-06700841
Description: Plasma decay half-life is the time measured for the plasma concentration of PF-06700841 to decrease by one half.
Time Frame: SAD: pre--dose, 0.5,1,2,4,6,8,12,16,24,36,48,72,96 hour post-dose on Day 1; MAD: pre--dose 0.5,1,2,4,6,8,12,24 hour post-dose on Day 10; MAD Psoriasis: pre--dose, 0.5,1,2,4,6,8,12,16,24 hours post-dose on Day 28
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 7 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5 | 12 | 12 | 12
hour | NA (NA) [0.500 to 2.00] — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 4.554 (1.8066) [0.500 to 1.00] | 3.848 (1.1587) [0.500 to 1.00] | 4.363 (2.4126) [0.500 to 1.02] | 7.519 (2.8236) [0.500 to 2.00] | 6.813 (1.9875) [0.500 to 2.00] | 5.928 (3.3336) [1.00 to 1.03] | 4.860 (1.9304) [1.00 to 1.00] | 10.67 (1.8440) [1.00 to 2.00] | 9.133 (2.2579) [1.00 to 2.00] | 7.458 (2.1595) [0.500 to 2.00] | 16.01 (31.584) [0.983 to 2.00] | 6.032 (1.7121) [1.00 to 2.00] | 6.155 (1.4408) [0.500 to 2.00] | 6.168 (1.2965) [0.500 to 2.00] | 5.848 (1.4383) [1.00 to 4.00]

37. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Mean Residence Time (MRT) of PF-06700841
Description: MRT= AUMCinf/AUCinf, where AUMCinf is the area under the first moment curve from time 0 extrapolated to infinite time, calculated using the linear/log trapezoidal method.
Time Frame: SAD: pre--dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post-dose on Day 1; MAD: pre--dose 0.5, 1, 2, 4, 6, 8, 12, 24 hour post--dose on Day 10; MAD Psoriasis: pre--dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hours post-dose on Day 28
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 7 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5
hour | NA (NA) — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 6.414 (46) | 5.169 (34) | 5.206 (44) | 7.277 (37) | 8.758 (29) | 7.191 (45) | 6.830 (38) | 10.35 (25) | 9.592 (22) | 9.025 (26) | 6.072 (92) | 8.534 (36)

38. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Apparent Volume of Distribution (Vz/F) of PF-06700841
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: SAD: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post-dose on Day 1; MAD: pre-dose 0.5, 1, 2, 4, 6, 8, 12, 24 hour post-dose on Day 10; MAD Psoriasis: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hours post-dose on Day 28
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 7 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5
liter | NA (NA) [0.500 to 2.00] — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 126.4 (26) [0.500 to 1.00] | 151.0 (18) [0.500 to 1.00] | 115.7 (16) [0.500 to 1.02] | 210.5 (45) [0.500 to 2.00] | 102.4 (27) [0.500 to 2.00] | 177.6 (30) [1.00 to 1.03] | 106.2 (12) [1.00 to 1.00] | 249.4 (45) [1.00 to 2.00] | 180.9 (30) [1.00 to 2.00] | 112.4 (18) [0.500 to 2.00] | 245.4 (206) [0.983 to 2.00] | 109.6 (18) [1.00 to 2.00]

39. Secondary Outcome: Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Apparent Clearance (CL/F) of PF-06700841
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Clearance obtained after oral dose is influenced by the fraction of the dose absorbed. CL/F =Dose of PF-06700841/AUCinf.
Time Frame: SAD: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hour post-dose on Day 1; MAD: pre-dose 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hour post-dose on Day 10; MAD Psoriasis: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hours post-dose on Day 28
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 7 | 8 | 5 | 3 | 6 | 4 | 4 | 7 | 5
Liter per hour (L/hr) | NA (NA) — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 20.57 (61) | 28.26 (31) | 20.82 (65) | 20.85 (61) | 10.86 (46) | 23.65 (41) | 15.95 (51) | 16.43 (38) | 14.03 (35) | 10.83 (16) | 30.30 (103) | 13.04 (43)

40. Secondary Outcome: Multiple Ascending Dose (MAD) and MAD Psoriasis Cohort: Peak-Trough Fluctuation (PTF) of PF-06700841
Description: PTF was calculated as: Cmax-Cmin/Cavg. Cmax is the maximum observed plasma concentration of PF-06700841. Cmin is the minimum observed plasma concentration of PF-06700841. Cavg is the average observed plasma concentration of PF-06700841 calculated as area under the plasma concentration-time curve during a dosing Interval (AUC[tau]) divided by the dosing interval (tau), where dosing interval was 24 hours for MAD once daily cohorts, 12 hours for MAD twice daily cohort and 24 hours for MAD Psoriasis cohort.
Time Frame: MAD: pre--dose 0.5, 1, 2, 4, 6, 8, 12, 24 hour post--dose on Day 10; MAD Psoriasis: pre--dose, 0.5,1,2,4,6,8,12,16,24 hours post-dose on Day 28
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 4 | 4 | 5
ratio | 2.815 (40) | 3.543 (38) | 2.643 (31) | 1.297 (22) | 2.911 (43) | 3.414 (44) | 2.654 (42)

41. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Amount of PF-06700841 Recovered Unchanged in the Urine Over the Time Interval Tau (Aetau)
Description: Aetau is the amount of drug recovered unchanged in urine during the dosing interval (tau), where dosing interval was 24 hours for MAD once daily cohorts, 12 hours for MAD twice daily cohort.
Time Frame: 0-24 hour on Day 10
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 5 | 3 | 1 | 4 | 4
milligram | 1.109 (45) | 2.798 (57) | NA (NA) — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 7.758 (57) | 15.60 (44)

42. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Percentage of Dose of PF-06700841 Recovered Unchanged in the Urine Over the Time Interval Tau (Aetau%)
Description: Aetau% was calculated as: 100*Aetau/dose. Aetau is the amount of drug recovered unchanged in urine during the dosing interval (tau), where dosing interval was 24 hours for MAD once daily cohorts, 12 hours for MAD twice daily cohort.
Time Frame: 0-24 hours on Day 10
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose recovered
Arm/Group | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 5 | 3 | 6 | 4 | 4
percentage of dose recovered | 11.09 (45) | 9.332 (57) | NA (NA) — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 15.54 (57) | 8.910 (44)

43. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Renal Clearance
Description: Renal clearance was calculated as amount of drug recovered unchanged in urine during the dosing interval tau (Aetau) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau), where dosing interval was 24 hours for MAD once daily cohorts, 12 hours for MAD twice daily cohort.
Time Frame: 0-24 hours on Day 10
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 5 | 3 | 1 | 4 | 4
Liter per hour | 2.619 (18) | 1.486 (15) | NA (NA) — Data was not collected due to less than 3 participants were evaluable and considered insufficient to calculate a reliable estimation, by investigator. | 2.179 (31) | 0.9629 (58)

44. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Interferon Gamma-induced Protein 10 (IP-10) Concentration in Serum at Baseline
Description: Serum samples for IP-10 were analyzed using a validated analytical assay. Lower limit of quantification (LLOQ) for IP-10 was 10 pg/mL.
Time Frame: Baseline
Population: Pharmacodynamic (PD) analysis set included all randomized and treated participants who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
picogram per milliliter (pg/mL) | 119.17 (40.090) | 188.76 (238.380) | 219.62 (275.440) | 78.28 (29.481) | 141.38 (100.403) | 115.00 (38.458) | 114.33 (26.164)

45. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Interferon Gamma-induced Protein 10 (IP-10) Concentration in Serum at Day 2, 5, 10, 11, 28
Description: Serum samples for IP-10 were analyzed using a validated analytical assay. LLOQ for IP-10 was 10 pg/mL.
Time Frame: Baseline, Day 2, 5, 10, 11, 28
Population: PD analysis set included all randomized and treated participants who had at least 1 of the PD parameters of. Here, 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
pg/mL
  Baseline (n =9, 2, 5, 4, 6, 5, 6) | 114.04 (70.658) | 85.50 (13.011) | 101.12 (56.853) | 142.23 (165.924) | 106.43 (28.244) | 121.60 (20.959) | 135.42 (57.855)
  Change at Day 2 (n =9, 2, 5, 4, 6, 5, 6) | 5.66 (13.421) | 2.00 (13.294) | -20.14 (41.966) | -23.60 (82.888) | -47.52 (19.664) | -60.64 (16.913) | -67.73 (35.998)
  Change at Day 5 (n =9, 2, 5, 4, 6, 5, 6) | 4.33 (12.213) | -3.25 (13.506) | -42.12 (48.250) | -53.40 (125.815) | -55.80 (15.273) | -71.40 (11.857) | -80.65 (66.445)
  Change at Day 10 (n =9, 2, 5, 3, 6, 4, 4) | -1.92 (24.123) | 4.75 (9.687) | -40.10 (43.129) | -96.67 (134.176) | -57.22 (9.321) | -70.50 (14.007) | -106.40 (60.163)
  Change at Day 11 (n =9, 2, 5, 3, 6, 4, 4) | 11.01 (19.008) | 1.85 (0.778) | -37.56 (47.031) | -102.53 (131.223) | -37.95 (24.957) | -54.25 (23.972) | -112.20 (60.459)
  Change at Day 28 (n =9, 2, 5, 3, 6, 4, 4) | -14.59 (21.736) | 2.85 (11.102) | -11.76 (51.955) | -62.07 (94.378) | 8.48 (23.010) | 18.30 (34.748) | -47.15 (89.356)

46. Secondary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Interferon Gamma-Induced Protein 10 (IP-10) Concentration in Serum at Day 2, 5, 7, 14, 21, 28, 29, 35, 56
Description: as for outcome 44
Time Frame: Baseline, Day 2, 5, 7, 14, 21, 28, 29, 35, 56
Population: PD analysis set included all randomized and treated participants who had at least 1 of the PD parameters of interest. Here, 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
pg/mL
  Baseline (n =9, 14, 7) | 302.00 (281.552) | 127.58 (45.829) | 123.09 (22.244)
  Change at Day 2 (n =9, 14, 7) | 53.44 (214.334) | -8.51 (34.704) | -49.57 (35.759)
  Change at Day 5 (n =9, 14, 7) | -21.63 (142.195) | -33.93 (33.465) | -49.01 (35.998)
  Change at Day 7 (n =9, 12, 7) | -25.71 (133.510) | -31.31 (32.203) | -52.50 (42.216)
  Change at Day 14 (n =9, 10, 6) | -69.91 (106.951) | -52.06 (24.663) | -68.55 (28.524)
  Change at Day 21 (n =9, 9, 5) | -42.87 (122.986) | -51.47 (28.094) | -46.64 (27.340)
  Change at Day 28 (n =8, 7, 5) | -1.0 (31.351) | -46.19 (35.893) | -53.36 (19.771)
  Change at Day 29 (n =8, 7, 5) | -22.20 (95.930) | -37.50 (31.849) | -49.34 (14.306)
  Change at Day 35 (n =8, 6, 5) | -69.54 (124.165) | 10.45 (37.860) | 110.68 (108.041)
  Change at Day 56 (n =7, 6, 4) | -31.71 (67.158) | 16.18 (19.348) | 167.85 (201.780)

47. Secondary Outcome: Single Ascending Dose (SAD) Cohort: High Sensitivity C-reactive Protein (hsCRP) Concentration in Serum at Baseline
Description: Serum samples for hsCRP were analyzed using a validated analytical assay. Reference range for measurement of CRP was 0.015 to 2.0 mg/dL. LLOQ for hsCRP was 0.03 mg/dL and limit of detection was 0.015 mg/dL.
Time Frame: Baseline
Population: PD analysis set included all randomized and treated participants who had at least 1 of the PD parameters of interest.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
milligram per deciliter (mg/dL) | 0.1220 (0.11909) | 0.1066 (0.09662) | 0.6420 (1.41413) | 0.0757 (0.04523) | 0.2290 (0.11714) | 0.1158 (0.20871) | 0.1710 (0.10387)

48. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline In High Sensitivity C-reactive Protein (hsCRP) at Day 2, 5, 10, 11, 28
Description: as for outcome 47
Time Frame: Baseline, Day 2, 5, 10, 11, 28
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
mg/dL
  Baseline (n= 9, 2, 5, 4, 6, 5, 6) | 0.0974 (0.06791) | 0.0815 (0.08556) | 0.1002 (0.11675) | 0.0983 (0.03734) | 0.0505 (0.02799) | 0.0746 (0.02523) | 0.1902 (0.06394)
  Change at Day 2 (n= 9, 2, 5, 4, 6, 5, 6) | -0.0148 (0.03176) | -0.0205 (0.00071) | -0.0670 (0.08196) | -0.0408 (0.03052) | -0.0212 (0.01712) | -0.0298 (0.01743) | -0.0307 (0.08168)
  Change at Day 5 (n= 9, 2, 5, 4, 6, 5, 6) | -0.0352 (0.03847) | -0.0050 (0.02263) | -0.0972 (0.11656) | -0.0753 (0.02269) | -0.0435 (0.02202) | -0.0596 (0.03345) | -0.1078 (0.05948)
  Change at Day 10 (n= 9, 2, 5, 3, 6, 4, 4) | -0.0329 (0.05656) | 0.0015 (0.00778) | -0.1002 (0.11675) | -0.0903 (0.00961) | -0.0467 (0.02881) | -0.0618 (0.01445) | -0.1838 (0.04529)
  Change at Day 11 (n= 9, 2, 5, 3, 6, 4, 4) | -0.0186 (0.07315) | -0.0040 (0.00990) | -0.1002 (0.11675) | -0.0870 (0.00819) | -0.0435 (0.02849) | -0.0615 (0.01330) | -0.1878 (0.04136)
  Change at Day 28 (n= 9, 2, 5, 3, 6, 4, 4) | 0.0496 (0.18748) | 0.0790 (0.08910) | -0.0352 (0.15033) | 0.0023 (0.06001) | 0.0223 (0.01556) | -0.0275 (0.04086) | 1.1255 (1.63253)

49. Secondary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline In High Sensitivity C-reactive Protein (hsCRP) at Day 2, 5, 7, 14, 21, 28, 29, 35 and 56
Description: as for outcome 47
Time Frame: Baseline, Day 2, 5 ,7,14, 21, 28, 29, 35, 56
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
mg/dL
  Baseline (n =9, 14, 7) | 1.0699 (1.39179) | 0.5694 (1.11752) | 0.3143 (0.34167)
  Change at Day 2 (n =9, 14, 7) | -0.1096 (0.25370) | -0.3408 (0.86901) | -0.0189 (0.14180)
  Change at Day 5 (n =9, 14, 7) | 0.0204 (0.51424) | -0.2413 (1.45363) | -0.2119 (0.27245)
  Change at Day 7 (n =9, 12, 7) | 0.1958 (0.85725) | -0.1573 (1.90640) | -0.1983 (0.31021)
  Change at Day 14 (n =9, 10, 6) | 0.4118 (1.19190) | -0.1910 (0.65215) | -0.2582 (0.33762)
  Change at Day 21 (n =9, 9, 5) | -0.1397 (0.46958) | -0.3067 (0.61035) | -0.2716 (0.38954)
  Change at Day 28 (n =8, 7, 5) | -0.4075 (0.37814) | -0.3549 (0.69576) | -0.2670 (0.37674)
  Change at Day 29 (n =8, 7, 5) | -0.6113 (0.79373) | -0.3533 (0.69589) | -0.2626 (0.34387)
  Change at Day 35 (n =8, 6, 5) | -0.5945 (0.78042) | -0.2533 (0.79446) | 0.7546 (1.07215)
  Change at Day 56 (n =7, 6, 4) | -0.3407 (0.45280) | -0.2662 (0.78307) | 0.2533 (0.82107)

50. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Neutrophil Counts at Day 2, 5 and 8
Time Frame: Baseline, Day 2, 5, 8
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: cells per millimeter cube (cells/mm^3)
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
cells per millimeter cube (cells/mm^3)
  Baseline (n =13, 7, 6, 6, 6, 8, 8) | 2.988 (1.2090) | 2.433 (1.0574) | 3.097 (1.1903) | 2.500 (0.6782) | 3.048 (0.7552) | 2.973 (1.2374) | 2.858 (0.6901)
  Change at Day 2 (n =13, 7, 6, 6, 6, 8, 8) | 0.096 (0.7459) | 0.340 (0.6643) | 0.377 (0.7133) | 0.285 (0.3214) | 0.240 (0.7344) | -0.315 (0.8594) | -0.760 (0.5266)
  Change at Day 5 (n =13, 6, 6, 6, 5, 8, 8) | 0.047 (0.8048) | 0.280 (0.5187) | -0.162 (1.1032) | -0.170 (0.2265) | -0.170 (0.6963) | 0.296 (0.3849) | 0.654 (0.6930)
  Change at Day 8 (n =12, 5, 6, 6, 5, 8, 8) | -0.245 (0.7834) | 0.196 (0.1674) | 0.017 (1.1173) | -0.293 (0.3100) | -0.058 (0.9051) | -0.110 (0.7910) | 1.188 (1.8134)

51. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Neutrophil Counts at Day 4, 8, 10, 11, 14, 28
Time Frame: Baseline, Day 4, 8, 10, 11, 14, 28
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
cells/mm^3
  Baseline (n =9, 2, 5, 4, 6, 5, 6) | 2.584 (0.8858) | 2.340 (0.2970) | 2.676 (0.6726) | 2.770 (0.4907) | 2.710 (1.0372) | 2.690 (0.9337) | 3.217 (0.9677)
  Change at Day 4 (n =9, 2, 5, 4, 6, 5, 6) | 0.099 (0.4191) | 0.060 (0.0283) | -0.242 (1.1533) | -0.215 (0.6376) | -0.295 (0.8000) | -0.980 (0.3726) | -0.902 (2.0680)
  Change at Day 8 (n =9, 2, 5, 4, 6, 4, 5) | 0.239 (0.5725) | 0.635 (1.1526) | -0.296 (0.7032) | -0.178 (0.5160) | -0.793 (0.5720) | -0.913 (0.4039) | -1.702 (1.3292)
  Change at Day 10 (n =9, 2, 5, 3, 6, 4, 4) | 0.156 (0.5860) | 0.635 (1.0394) | -0.340 (0.8602) | 0.327 (0.8228) | -1.012 (0.5365) | -1.168 (0.4197) | -2.125 (1.2878)
  Change at Day 11 (n =9, 2, 5, 3, 6, 4, 4) | 0.158 (0.4996) | 0.400 (1.2021) | -0.382 (0.8244) | 0.260 (0.7572) | -0.280 (0.9159) | -0.248 (0.3976) | -2.010 (1.3075)
  Change at Day 14 (n =9, 2, 5, 3, 6, 4, 4) | -0.020 (0.5471) | 0.385 (0.8273) | -0.060 (0.8663) | 0.650 (0.8543) | 0.232 (0.4395) | 0.228 (0.3377) | 0.290 (1.0943)
  Change at Day 28 (n =9, 2, 5, 3, 6, 4, 4) | 0.030 (0.4649) | 0.130 (0.4525) | -0.012 (1.1401) | 0.697 (0.0839) | -0.055 (0.4578) | 0.050 (0.6249) | 0.298 (0.3777)

52. Secondary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Neutrophil Counts at Day 4, 6, 8, 10, 13, 14, 21, 28, 35, 42 and 56
Time Frame: Baseline, Day 4, 6 ,8,10, 13, 14, 21, 28, 35, 42, 56
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
cells/mm^3
  Baseline (n =9, 14, 7) | 4.109 (1.4401) | 3.640 (1.4997) | 3.909 (1.1841)
  Change at Day 4 (n =9, 14, 7) | -0.402 (0.9308) | 0.006 (1.1696) | 0.153 (0.7114)
  Change at Day 6 (n =9, 14, 7) | -0.209 (1.2224) | -0.073 (0.8229) | -0.303 (0.6058)
  Change at Day 8 (n =9, 12, 7) | -0.473 (0.6962) | 0.013 (1.2572) | -0.973 (0.4394)
  Change at Day 10 (n =9, 10, 7) | -0.463 (0.7834) | 0.197 (1.1099) | -1.299 (0.6906)
  Change at Day 13 (n =9, 10, 6) | -0.654 (0.7847) | -0.297 (1.2264) | -1.538 (0.9097)
  Change at Day 14 (n =9, 10, 6) | -0.247 (0.9682) | -0.146 (1.1226) | -1.465 (0.9517)
  Change at Day 21 (n =9, 9, 5) | -0.762 (0.7389) | -0.638 (0.9404) | -1.410 (1.2572)
  Change at Day 28 (n =8, 7, 5) | -0.678 (0.6416) | -0.890 (0.9952) | -1.450 (1.1195)
  Change at Day 35 (n =8, 6, 5) | -0.081 (1.4496) | -0.777 (1.1154) | -1.008 (0.8082)
  Change at Day 42 (n =7, 6, 4) | -0.427 (0.6004) | -0.677 (1.1209) | -1.050 (0.6868)
  Change at Day 56 (n =7, 6, 4) | -0.036 (0.7864) | -0.533 (1.3025) | -0.493 (1.6373)

53. Secondary Outcome: Single Ascending Dose (SAD) Cohort: Change From Baseline in Reticulocyte Counts at Day 2, 5, 8
Time Frame: Baseline, Day 2, 5, 8
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo: SAD Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 200 mg SAD Cohort
Number analyzed (Participants) | 13 | 7 | 6 | 6 | 6 | 8 | 8
cells/mm^3
  Baseline (n =13, 7, 6, 6, 6, 8, 8) | 1.23 (0.470) | 1.19 (0.380) | 0.98 (0.279) | 1.25 (0.243) | 1.25 (0.327) | 1.44 (0.825) | 1.20 (0.524)
  Change at Day 2 (n =13, 7, 6, 6, 6, 8, 8) | 0.02 (0.152) | -0.09 (0.135) | -0.02 (0.160) | -0.15 (0.138) | 0.02 (0.256) | -0.14 (0.177) | -0.16 (0.177)
  Change at Day 5 (n =13, 6, 6, 6, 5, 8, 8) | 0.04 (0.194) | 0.07 (0.175) | -0.05 (0.138) | -0.27 (0.103) | 0.02 (0.409) | -0.23 (0.459) | -0.15 (0.193)
  Change at Day 8 (n =12, 5, 6, 6, 5, 8, 8) | 0.03 (0.234) | 0.04 (0.114) | 0.03 (0.242) | -0.15 (0.226) | 0.34 (0.532) | -0.26 (0.478) | -0.14 (0.346)

54. Secondary Outcome: Multiple Ascending Dose (MAD) Cohort: Change From Baseline in Reticulocyte Counts at Day 4, 8, 10, 11, 14 and 28
Time Frame: Baseline, Day 4, 8, 10, 11, 14, 28
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort
Number analyzed (Participants) | 9 | 2 | 5 | 4 | 6 | 5 | 6
cells/mm^3
  Baseline (n =9, 2, 5, 4, 6, 5, 6) | 1.26 (0.490) | 0.85 (0.212) | 1.22 (0.363) | 1.03 (0.350) | 1.40 (0.410) | 2.26 (0.550) | 1.38 (0.286)
  Change at Day 4 (n =9, 2, 5, 4, 6, 5, 6) | -0.03 (0.212) | 0.05 (0.071) | -0.10 (0.071) | 0.05 (0.129) | -0.18 (0.306) | -0.54 (0.241) | -0.32 (0.223)
  Change at Day 8 (n =9, 2, 5, 4, 6, 4, 5) | -0.11 (0.285) | 0.30 (0.283) | -0.20 (0.100) | -0.13 (0.250) | -0.60 (0.210) | -1.28 (0.395) | -0.90 (0.187)
  Change at Day 10 (n =9, 2, 5, 3, 6, 4, 4) | -0.19 (0.398) | 0.20 (0.283) | -0.24 (0.089) | -0.07 (0.231) | -0.70 (0.352) | -1.48 (0.403) | -0.93 (0.206)
  Change at Day 11 (n =9, 2, 5, 3, 6, 4, 4) | -0.13 (0.343) | 0.30 (0.424) | -0.34 (0.089) | -0.23 (0.115) | -0.72 (0.354) | -1.43 (0.499) | -0.93 (0.330)
  Change at Day 14 (n =9, 2, 5, 3, 6, 4, 4) | -0.12 (0.393) | 0.05 (0.495) | -0.22 (0.110) | 0.03 (0.058) | -0.60 (0.297) | -1.10 (0.408) | -0.90 (0.183)
  Change at Day 28 (n =9, 2, 5, 3, 6, 4, 4) | 0.11 (0.431) | -0.05 (0.212) | 0.22 (0.277) | 0.30 (0.346) | 0.65 (0.619) | 0.18 (0.189) | 0.33 (0.479)

55. Secondary Outcome: Multiple Ascending Dose (MAD) Psoriasis Cohort: Change From Baseline in Reticulocyte Counts at Day 4, 6, 8, 10, 13, 14, 21, 28, 35, 42 and 56
Time Frame: Baseline, Day 4, 6 ,8,10, 13, 14, 21, 28, 35, 42, 56
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Placebo: MAD Psoriasis Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort
Number analyzed (Participants) | 9 | 14 | 7
cells/mm^3
  Baseline (n =9, 14, 7) | 1.49 (0.355) | 1.45 (0.285) | 1.31 (0.393)
  Change at Day 4 (n =9, 14, 7) | -0.10 (0.300) | -0.09 (0.207) | -0.13 (0.281)
  Change at Day 6 (n =9, 14, 7) | -0.09 (0.392) | -0.16 (0.250) | -0.27 (0.373)
  Change at Day 8 (n =9, 12, 7) | -0.20 (0.430) | -0.21 (0.243) | -0.59 (0.353)
  Change at Day 10 (n =9, 10, 7) | -0.21 (0.355) | -0.35 (0.295) | -0.70 (0.361)
  Change at Day 13 (n =9, 10, 6) | -0.20 (0.354) | -0.41 (0.373) | -0.75 (0.459)
  Change at Day 14 (n =9, 10, 6) | -0.13 (0.371) | -0.34 (0.392) | -0.82 (0.462)
  Change at Day 21 (n =9, 9, 5) | -0.22 (0.393) | -0.27 (0.430) | -0.66 (0.270)
  Change at Day 28 (n =8, 7, 5) | -0.24 (0.487) | -0.36 (0.264) | -0.60 (0.255)
  Change at Day 35 (n =8, 6, 5) | 0.26 (0.498) | -0.03 (0.163) | 0.22 (0.228)
  Change at Day 42 (n =7, 6, 4) | 0.46 (0.431) | 0.33 (0.427) | 1.35 (0.551)
  Change at Day 56 (n =7, 6, 4 | 0.13 (0.335) | 0.07 (0.250) | 0.50 (0.183)

ADVERSE EVENTS:
Arm/Group | Placebo: SAD Cohort | Placebo: Once Daily MAD Cohort | Placebo: Twice Daily MAD Cohort | Placebo: MAD Psoriasis Cohort | PF--06700841: 1 Milligram (mg) SAD Cohort | PF--06700841: 3 mg SAD Cohort | PF-06700841: 10 mg SAD Cohort | PF-06700841: 10 mg Once Daily MAD Cohort | PF-06700841: 30 mg SAD Cohort | PF-06700841: 30 mg Once Daily MAD Cohort | PF-06700841: 100 mg SAD Cohort | PF-06700841: 100 mg Once Daily MAD Cohort | PF-06700841: 50 mg Twice Daily MAD Cohort | PF-06700841: 200 mg SAD Cohort | PF-06700841: 175 mg Once Daily MAD Cohort | PF-06700841: 30 mg MAD Psoriasis Cohort | PF-06700841: 100 mg MAD Psoriasis Cohort | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9 | 0/2 | 0/9 | 0/7 | 0/6 | 0/6 | 0/5 | 0/6 | 0/4 | 0/8 | 0/6 | 0/5 | 0/8 | 0/6 | 0/14 | 0/7 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/13 | 0/9 | 1/2 | 5/9 | 1/7 | 1/6 | 0/6 | 3/5 | 1/6 | 2/4 | 3/8 | 3/6 | 5/5 | 2/8 | 5/6 | 11/14 | 6/7 | 1/12 | 2/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: SAD Cohort (N=13) | Placebo: Once Daily MAD Cohort (N=9) | Placebo: Twice Daily MAD Cohort (N=2) | Placebo: MAD Psoriasis Cohort (N=9) | PF--06700841: 1 Milligram (mg) SAD Cohort (N=7) | PF--06700841: 3 mg SAD Cohort (N=6) | PF-06700841: 10 mg SAD Cohort (N=6) | PF-06700841: 10 mg Once Daily MAD Cohort (N=5) | PF-06700841: 30 mg SAD Cohort (N=6) | PF-06700841: 30 mg Once Daily MAD Cohort (N=4) | PF-06700841: 100 mg SAD Cohort (N=8) | PF-06700841: 100 mg Once Daily MAD Cohort (N=6) | PF-06700841: 50 mg Twice Daily MAD Cohort (N=5) | PF-06700841: 200 mg SAD Cohort (N=8) | PF-06700841: 175 mg Once Daily MAD Cohort (N=6) | PF-06700841: 30 mg MAD Psoriasis Cohort (N=14) | PF-06700841: 100 mg MAD Psoriasis Cohort (N=7) | PF-06700841: 100 mg Tab Fasted (Food Effect Cohort) (N=12) | PF-06700841: 100 mg Solution Fasted (Food Effect Cohort) (N=12) | PF-06700841: 100 mg Tablet Fed (Food Effect Cohort) (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4 | 1 | 4 | 7 | 6 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.